CLINICAL TRIAL: NCT02305654
Title: International Penile Advanced Cancer Trial (International Rare Cancers Initiative Study)
Acronym: InPACT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: National Cancer Institute (NCI) (NIH); ECOG-ACRIN Cancer Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR CTSU/2014/10048; CRUK/13/005 (Other Grant/Funding Number: Cancer Research UK); 13580965 (Registry Identifier: ISRCTN); EA8134 (Other Grant/Funding Number: NCI); IRCI004 (Other: IRCI); 2015-001199-23 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-12-02 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of the Penis, Usual Type
Keywords: Penis cancer; Chemotherapy; Chemoradiotherapy; Surgery; Phase III
MeSH Terms: conditions — Penile Neoplasms | interventions — Paclitaxel; Ifosfamide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm A - Standard Surgery (ILND) (Active Comparator): Part of randomisation 1.
  The total treatment duration (Inguinal Lymph Node Dissection (ILND)) is estimated to be over 1 day for those patients allocated to Arm A - standard surgery.
  Interventions: Procedure: ILND - Inguinal Lymph Node Dissection
- Arm B - neoadjuvant chemotherapy (Experimental): Part of randomisation 1.
  Patients will receive up to 4 cycles of Paclitaxel, Ifosfamide, and Cisplatin (TIP).
  Administration on an outpatient basis:
  Paclitaxel 175 mg/m2, day 1, Ifosfamide 900 mg/m2, days 2-5, Cisplatin 15 mg/m2, days 1-5
  Administration on an inpatient basis:
  Paclitaxel 175 mg/m2, day 1, Ifosfamide 1200 mg/m2, days 1-3, Cisplatin 25 mg/m2, days 1-3
  Interventions: Drug: Paclitaxel; Drug: Ifosfamide; Drug: Cisplatin
- Arm C - neoadjuvant chemoradiotherapy (Experimental): Part of randomisation 1.
  Radiotherapy dose is 45Gy in 25 fractions over 5 weeks using 6-10 MV photons to all regions.
  Concurrent cisplatin 40mg/m2 will be given weekly, subject to GFR>45mls/min.
  Interventions: Drug: Cisplatin; Radiation: Intensity modulated radiation treatment (IMRT)
- Arm P - prophylactic PLND (Experimental): Part of randomisation 2.
  Prophylactic pelvic lymph node dissection (PLND) - The total treatment duration is estimated to be over 1 day.
  Patients who have NOT received neoadjuvant chemoradiotherapy will receive adjuvant chemoradiotherapy:
  Cisplatin 40mg/m2 will be given weekly, subject to GFR>45mls/min.
  Groin: One or both groins may be boosted up to 54Gy in 25 fractions. An IMRT boost of up to 57 Gy can be given to recurrent or residual macroscopic tumour
  Pelvis: the dose is limited to 45Gy unless IMRT is available. An IMRT boost of up to 54Gy in 25 fractions is applied to:
  1. Any macroscopic tumour or pathological lymph nodes
  2. Electively to external iliac nodes in patient with high disease burden
  Patients who have had neoadjuvant chemoradiotherapy will have prophylactic PLND alone.
  Interventions: Procedure: Prophylactic PLND - pelvic lymph node dissection
- Arm Q - Surveillance no prophylactic PLND (No Intervention): no prophylactic PLND Part of randomisation 2.
  For patients who have NOT received neoadjuvant chemoradiotherapy:
  Groin: One or both groins may be boosted up to 54Gy in 25 fractions. An IMRT boost of up to 57 Gy can be given to recurrent or residual macroscopic tumour
  Pelvis: the dose is limited to 45Gy unless IMRT is available. An IMRT boost of up to 54Gy in 25 fractions is applied to:
  Any macroscopic tumour or pathological lymph nodes Electively to external iliac nodes in patient with high disease burden

INTERVENTIONS:
Procedure: ILND - Inguinal Lymph Node Dissection — Surgery to remove the lymph nodes in the groin near to where the cancer first appeared.
  Arms: Arm A - Standard Surgery (ILND)
Drug: Paclitaxel — Dose 175mg/m2 as part of TIP regimen.
  Other Names: Taxol
  Arms: Arm B - neoadjuvant chemotherapy
Drug: Ifosfamide — Dose 900mg/m2 as part of TIP regimen.
  Other Names: Mitoxana
  Arms: Arm B - neoadjuvant chemotherapy
Drug: Cisplatin — Dose 15mg/m2 as part of TIP regimen (neoadjuvant chemotherapy arm) Dose 40mg/m2 for use concurrently with raditotherapy (chemoradiotherapy arm)
  Arms: Arm B - neoadjuvant chemotherapy; Arm C - neoadjuvant chemoradiotherapy
Radiation: Intensity modulated radiation treatment (IMRT) — Treatment with very high energy X-rays (radiotherapy).
  Arms: Arm C - neoadjuvant chemoradiotherapy
Procedure: Prophylactic PLND - pelvic lymph node dissection — Surgery to remove the lymph nodes deeper in the pelvis, further away from where the cancer first appeared, that are at high risk of harbouring cancer.
  Arms: Arm P - prophylactic PLND

SUMMARY:
This is an international phase III trial, with a Bayesian design, incorporating two sequential randomisations. It efficiently examines a series of questions that routinely arise in the sequencing of treatment. The study design has evolved from lengthy international consultation that has enabled us to build consensus over which questions arise from current knowledge and practice. It will enable potential randomisation for the majority of patients with inguinal lymph node metastases and will provide data to inform future clinical decisions.

InPACT-neoadjuvant patients are stratified by disease burden as assessed by radiological criteria. Treatment options are then defined according to the disease burden strata. Treatment is allocated by randomisation. Patients may be allocated to one of three initial treatments:

A. standard surgery (ILND); B. neoadjuvant chemotherapy followed by standard surgery (ILND); or C. neoadjuvant chemoradiotherapy followed by standard surgery (ILND).

After ILND, patients are defined as being at low or high risk of recurrence based on histological interpretation of the ILND specimen. Patients at high risk of relapse are eligible for InPACT-pelvis, where they are randomised to either:

P. prophylactic PLND Q. no prophylactic PLND

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Measurable disease as determined by RECIST (version 1.1) criteria;
3. Histologically-proven squamous cell carcinoma of the penis,
4. Stage:

   * any T, N1 (i.e. a palpable mobile unilateral inguinal lymph node), M0 or;
   * any T, N2 (i.e. palpable mobile multiple or bilateral inguinal lymph nodes), M0 or;
   * any T, N3 (i.e. fixed inguinal nodal mass or any pelvic lymphadenopathy), M0
5. Performance Status ECOG 0, 1 or 2.

Exclusion Criteria:

1. Pure verrucous carcinoma of the penis,
2. Nonsquamous malignancy of the penis,
3. Squamous carcinoma of the urethra,
4. Stage M1,
5. Previous chemotherapy or chemoradiotherapy,
6. Concurrent malignancy (other than SCC or Basal Cell Carcinoma of non-penile skin) that has required surgical or non-surgical treatment in the last 3 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 5 years
  The primary outcome measure that will be measured for all trial patients is survival time. This is defined in whole days as the time from the date of randomisation to the date of death from any cause; for those who have not been reported as dead at the time of analysis, the survival time will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Disease specific survival time | up to 5 years
  Disease-specific survival time which is defined in whole days as the time from the date of randomisation to the date of death specifically from disease; for those who have not been reported as dead at the time of analysis, the survival time will be censored at the date of last follow-up and for those whose death is reported as non-disease specific then the survival time will be censored at date of death.
Number of patients experience a grade 3 or 4 toxicity | up to 5 years
Disease-free survival time | up to 5 years
  Disease-free survival time (DFST) which is defined in whole days as the time from date of randomisation to the date of either locoregional recurrence, distant metastasis or death from disease, whichever occurs first; for those who have not been reported as experiencing any of these events, the DFST will be censored at the date last known to be alive and free of disease or date of non-disease-specific death. A supplementary exploratory outcome measure will also be calculated taking date of penectomy as the origin rather than date of randomisation.
  Subsidiary outcome measures will be
  * locoregional recurrence free survival time (LRFST).
  * distant metastases free survival time (DMFST).
  * A supplementary exploratory outcome measure will also be calculated taking date of penectomy as the origin for all these outcome measures rather than date of randomisation.
Occurrence of surgical complication | up to 5 years
Is it possible to achieve pathological nodal assessment after chemotherapy | 12 weeks
  Feasibility of pathological nodal assessment after chemotherapy which is recorded as whether or not it was possible to achieve a pathological nodal assessment after chemotherapy.
Quality of life | Baseline, 3, 6, 9, 12, 18, 24 and 36 months
  Measured using the EORTC-QLQC30 and Lymphodema-QL
Occurrence of Pathological complete remission | Time to complete remission after randomisation
  Measured for all patients in InPACT-neoadjuvant:
  Absolute absence of disease on histological examination
Operability | 2-6 weeks
  Measured for all trial patients in InPACT-neoadjuvant. Operability which will be recorded as whether or not the planned inguinal node dissection was undertaken and the reasons if it did not occur.
Occurrence of Lower limb/scrotal oedema | up to 5 years
  Occurrence of Lower limb/scrotal oedema which is recorded as whether or not the patient experiences a lower limb or scrotal oedema
On-schedule delivery of neoadjuvant therapy | After randomisation up to 12 weeks
  Feasibility of on-schedule delivery of neoadjuvant therapy

OTHER OUTCOMES:
Acceptability of randomisation | up to 5 years
  In addition to the outcome measures, the acceptability of both randomisations will be monitored based on the proportion of eligible patients approached for randomisation, the proportion of approached patients consenting to randomisation and the proportion of randomised patients receiving their allocated treatment. This will provide ongoing information regarding the feasibility of the trial successfully completing to target.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Nicholson, Study Chair — Mid and South Essex NHS Foundation Trust; Curtis Pettaway, Study Chair — University of Texas M.D. Anderson Cancer Center ; 713-792-3250 ; cpettawa@mdanderson.org
Locations (17):
- United States (11):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- United Kingdom (6):
  - Velindre NHS Trust, Cardiff
  - University Hospitals of Leicester NHS Trust, Leicester
  - The Royal Marsden NHS Foundation Trust, London
  - St George's Hospital NHS Foundation Trust, London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.icr.ac.uk/our-research/our-research-centres/clinical-trials-and-statistics-unit/clinical-trials/inpact